CLINICAL TRIAL: NCT00738153
Title: Efficacy and Safety Study of Levemir® (Insulin Detemir) to Treat Type 1 and 2 Diabetes Mellitus
Brief Title: An Observational Study on Efficacy and Safety in Subjects Using Levemir® for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3536
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Levemir®

SUMMARY:
This observational study is conducted in Africa. The aim of this observational study is to evaluate the efficacy and the incidence of serious adverse drug reactions while using insulin Levemir® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with Type 1 or Type 2 diabetes mellitus is eligible for the study, including newly-diagnosed subjects who have never received insulin or an insulin analogue before. The selection of the subjects will be at the discretion of the individual physician

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for the final visit
* Currently being treated with insulin detemir
* Previously enrolled in this study
* Hypersensitivity to insulin detemir or to any of the excipients
* Pregnancy, breast-feeding, the intention to become pregnant or judged not to be using adequate contraceptive measures.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 1 or type 2 diabetes is eligible for the study, including newly-diagnosed subjects who have never received insulin or an insulin analogue before
Sampling Method: Non-Probability Sample
Enrollment: 798 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The incidence of serious adverse drug reactions, including major hypoglycaemic events | From baseline to 12 and 24 weeks of Levemir® therapy, respectively

SECONDARY OUTCOMES:
Number of serious adverse events | From baseline to 12 and 24 weeks of Levemir® therapy, respectively
Number of all adverse events | From baseline to 12 and 24 weeks of Levemir® therapy, respectively
Number of all hypoglycaemic events | in the 4 weeks preceding the visits at 12 weeks and 24 weeks.
Weight changes | at the end of study
HbA1c | at the end of study
Sub -group analysis of hypo risk | From baseline to 12 and 24 weeks of Levemir® therapy, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Casablanca, Morocco

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com